CLINICAL TRIAL: NCT01954277
Title: Immune-Pineal Axis Function in Chronic Tension-Type Headache: Noradrenergic Modulation and the Effect of Electroacupuncture
Brief Title: Immune-Pineal Axis Function in Chronic Tension-Type Headache
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Wolnei Caumo, MD, PhD, Professor and coordinator of Pain & Neuromodulation Lab, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 09-259
Record Dates: First submitted 2013-09-15; First posted 2013-10-01 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Tension-Type Headache
Keywords: Chronic Tension-Type Headache; Electroacupuncture; Headache Impact; BDNF; TNF
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroacupuncture (Experimental): All patients will receive 10 electroacupuncture sessions.
  Interventions: Device: Electroacupuncture
- Placebo Sham (Sham Comparator): All patients will receive 10 placebo sham sessions.
  Interventions: Device: Placebo Sham

INTERVENTIONS:
Device: Electroacupuncture — Eletroacupuncture performed using acupuncture needles.
  Other Names: Electrical acupuncture
  Arms: Electroacupuncture
Device: Placebo Sham — Placebo Sham is performed using electrodes, without electrical stimulation. Lights and sounds were identical to active treatment.
  Other Names: Placebo; Sham
  Arms: Placebo Sham

SUMMARY:
The purpose of this study is to determine whether electroacupuncture is effective in the treatment of chronic tension-type headache, measured by Headache Impact Test, Visual Analogue Scale and biomarkers.

DETAILED DESCRIPTION:
Tension-type headache can be defined as a constant sensation of pressure or heaviness, and is a highly-prevalent condition in the health services. The objective of the present study is to investigate the function of the immuno-pineal axis in chronic tension headache, focussed on the neuro-immune regulatory dysfunction. In addition, the effect of neuro-stimulation (electroacupuncture) on the function of this axis will also be studied.

This is a clinical Trial study, randomised, in parallel, cross-over with a blinded assessor, and with a sham placebo control.

The study will be carried out in the Clinical Research Outpatient Clinic of the Hospital de Clínicas de Porto Alegre (HCPA), with women aged between 18 and 60 years old. The participants will respond to questionnaires at the beginning and end of each therapeutic intervention, with 24-hour urine, blood and saliva collection. The therapeutic intervention will include: 10 electroacupuncture sessions and 10 sham placebo sessions. The measurements taken will be: quality of life, depression, impact of headache on daily life, sleep quality, chronotropic types, immuno-inflammatory mediators, levels of 6-sulfatoxymelatonin, and salivary cortisol.

Through these interventions it is hoped that patients will present an improvement in their pain presentation, quality of life and sleep, as well as central autonomic regulation. Evidence for these hypotheses will support a minimally-invasive treatment, with few side-effects and a low cost.

ELIGIBILITY:
Inclusion Criteria:

* Women,
* Aged between 18 and 60 years old,
* Providing informed consent to participate in the study,
* Literate,
* Clinical diagnosis of Chronic Tension-Type Headache according to the International Headache Society.

Exclusion Criteria:

* Psychiatric or neurologic disorder that unable patient to consent and follow study protocol,
* De-compensated systemic disease,
* Chronic inflammatory disease (e.g. Systemic Lupus Erythematous, Rheumatoid Arthritis),
* HIV.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | An expected average of 3 months. (At baseline and at the end of each intervention period).
  The intensity of pain was measured by a 10 cm VAS. The scores range from no pain (zero) to the worst possible pain (10 cm).

SECONDARY OUTCOMES:
Headache Impact Test (HIT-6) | An expected average of 3 months. (At baseline and at the end of each intervention period).
  This test was developed in 2004, and has equivalent psychometric properties in nine languages, including Portuguese. It consists of six questions that assess the impact of headache on the ability to work, study, home and in social situations.

OTHER OUTCOMES:
Biomarkers (BDNF nd TNF) | An expected average of 3 months. (At baseline and at the end of each intervention period).
  The BDNF and the TNF will be measured by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD, PhD, Study Chair — Hospital de Clinicas de Porto Alegre; Mônica Chassot, Principal Investigator — Federal University of Health Science of Porto Alegre; Francislea C. Sehn, Principal Investigator — Federal University of Health Science of Porto Alegre; Rafael Vercelino, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (1):
- Hospital de Clinicas e Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil